CLINICAL TRIAL: NCT05890703
Title: Painless Sharp Wound Debridement With Lidocaine-23%-Tetra-caine-7% Gel Versus EMLA 5% Cream: a Single-blind, Crossover, Randomised, Controlled Trial
Brief Title: Painless Sharp Wound Debridement With Lidocaine-23%-Tetra-caine-7% Gel Versus EMLA 5% Cream
Acronym: LIDOTETRA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Juerg Hafner (Other)
Responsible Party: Sponsor-Investigator, Juerg Hafner, University Hospital Zurich, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LIDOTETRA
Record Dates: First submitted 2023-05-17; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Ulcus Cruris; Ecthyma; Ulcer, Leg; Ulcer Venous
Keywords: EMLA; Lidocain; Tetracain; Leg ulcer; Sharp Wound Debridement; Anesthesia
MeSH Terms: conditions — Foot Ulcer; Ecthyma; Leg Ulcer; Varicose Ulcer | interventions — IGF2BP2 protein, human; signal peptide peptidase; Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IMP2 (lidocaine-23%-tetracaine-7% gel) (Experimental)
  Interventions: Drug: IMP2 (lidocaine-23%-tetracaine-7% gel)
- IMP1 (EMLA 5% cream) (Active Comparator)
  Interventions: Drug: IMP1 (EMLA 5% cream)

INTERVENTIONS:
Drug: IMP2 (lidocaine-23%-tetracaine-7% gel) — Applied in a 2 mm thick even layer for 30 minutes on the ulcer with an occlusive dressing. During the second treatment the same dose is applied. Immediately after removal of the occlusive dressing, the rest of the preparation will be removed and sharp debridement will be performed. In order to minimise bias in this crossover trial, the localisation of start (most distal part of Wound) of sharp debridement and the sequence of sharp debridement (if more than one wound; from the largest to the smallest) is defined in the first visit.
  Arms: IMP2 (lidocaine-23%-tetracaine-7% gel)
Drug: IMP1 (EMLA 5% cream) — Applied in a 2 mm thick even layer for 30 minutes on the ulcer with an occlusive dressing. During the second treatment the same dose is applied. Immediately after removal of the occlusive dressing, the rest of the preparation will be removed and sharp debridement will be performed. In order to minimise bias in this crossover trial, the localisation of start (most distal part of Wound) of sharp debridement and the sequence of sharp debridement (if more than one wound; from the largest to the smallest) is defined in the first visit.
  Arms: IMP1 (EMLA 5% cream)

SUMMARY:
In a single-blind, crossover, randomized, controlled trial with 40 participants we aim to demonstrate superior anaesthetic efficacy of lidocaine-23%-tetracaine-7% (IMP2) gel over EMLA 5% cream (IMP1) at comparable safety in sharp wound debridement of chronic leg ulcers.

This is a monocentric investigator initiated trial conducted in the University Hospital Zurich.

In this longitudinal trial, participants receive a sequence of different treatments (treatments on different days) and therefore are randomly assigned to one of two treatment sequences. One-half of participants will first receive IMP1 (first treatment visit, randomized) and then IMP2 (second treatment visit, crossover); the other half of participants the reverse sequence (first treatment visit: IMP2, second treatment visit: IMP1).

Primary Objective: We want to show that IMP 2 (lidocaine-23%-tetracaine-7% gel) is more effective in pain reduction than IMP 1 (EMLA® 5% cream) in sharp wound debridement.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 18 years and 90 years
* Chronic leg ulcer(s) (duration > 4 weeks) with biofilm or necrotic layers which require consecutive sharp debridement for at least two times (of the same ulcer)
* Minimal ulcer area of 1 cm2
* Leg ulcer has to enter into one of the following well defined aetiologies: venous, mixed venous-arterial, arterial, hypertensive ischemic leg ulcer (Martorell), vasculitic, ecthyma (covering >90% of all observed leg ulcers)
* Informed consent as documented by signature and being able to follow the study protocol (cognition)
* Proficiency in German, oral and written information

Exclusion Criteria:

* Women who are pregnant or breastfeeding (Women of childbearing potential need to perform a pregnancy test (urine test) within 24 hours prior to the study intervention and need at least one simple acceptable contraceptive method)
* Participants with hypersensitivity or allergy to lidocaine, prilocaine, tetracaine or auxiliary supplies contained in either EMLA® 5% cream or lidocaine-23%-tetracaine-7% gel.
* Participants with peripheral neuropathy (over 4/10 insensitive points with Semmes monofilament) are excluded due to disturbed pain perception, which could potentially influence the results.
* Participants that were previously included in this clinical trial
* Participants with a total wound area larger than 200 cm2

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Local anaesthetic efficacy | 15 seconds after start of sharp debridement, pain will be assessed with Visual Analogue Scale
  Local anaesthetic efficacy during sharp wound debridement will be assessed with Visual Analogue Scale for pain 15 seconds after start of sharp debridement or earlier in case debridement is completed in less than 15 seconds or early terminated due to intolerable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, University Hospital of Zurich, Switzerland, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No